CLINICAL TRIAL: NCT02106156
Title: Noninterventional Study on the Quality Assurance of the Therapy of Chronic Hepatitis C With Peg-(40kd)-Interferon Alfa-2a (Pegasys®) and Ribavirin (e.g. Copegus®) With Main Focus Gastroenterologists - a Project in BNG (Association of German Resident Gastroenterologists), Part III
Brief Title: Observational Study Evaluating the Quality of Pegylated Interferon Alfa-2a and Ribavirin Treatment for Chronic Hepatitis C in Cooperation With the BNG (Association of German Resident Gastroenterologists)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21645
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Hepatitis C: Participants with chronic hepatitis C planned for treatment with peginterferon alfa-2a alone or in combination with ribavirin according to routine clinical practice will be observed in this study.
  Interventions: Drug: Pegylated interferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — Pegylated interferon alfa-2a administered according to corresponding summary of product characteristics (SmPC).
  Other Names: Pegasys®
Drug: Ribavirin — Ribavirin administered according to corresponding summary of product characteristics (SmPC).
  Other Names: Copegus®

SUMMARY:
This observational study will examine the efficacy and safety of pegylated interferon (peginterferon) alfa-2a, mostly in combination with ribavirin treatment in chronic hepatitis C (CHC). Quality of care will also be assessed. Approximately 12% of the interferon-treated CHC patient population in Germany is expected to be studied over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* Clinically diagnosed CHC with detectable virus replication
* Women of childbearing potential should use adequate contraception. It is important that female participants of childbearing potential and their sexual partners use 2 contraceptive methods at the same time during treatment and 4 months after treatment discontinuation. During this time pregnancy tests have to be performed monthly. Particular attention is also required and pregnancy should be avoided 7 months after treatment discontinuation in female sexual partners of male participants taking ribavirin (Copegus®). Both should use adequate contraception.

Exclusion Criteria:

* Any contraindications for peginterferon alfa-2a or ribavirin treatment
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CHC treated with peginterferon alfa-2a and ribavirin according to routine clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 10228 (Actual)
Dates: Start 2008-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Herne, Germany

REFERENCES:
- [Derived] Niederau C, Mauss S, Schober A, Stoehr A, Zimmermann T, Waizmann M, Moog G, Pape S, Weber B, Isernhagen K, Sandow P, Bokemeyer B, Alshuth U, Steffens H, Huppe D. Predictive factors for sustained virological response after treatment with pegylated interferon alpha-2a and ribavirin in patients infected with HCV genotypes 2 and 3. PLoS One. 2014 Sep 19;9(9):e107592. doi: 10.1371/journal.pone.0107592. eCollection 2014. PMID 25238535

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol participants were not allocated to study arms. Separation of participants was performed post hoc for all analyses. Participants who underwent elastography were allocated to separate arms as another time schedule was used and also untreated participants were documented, who were analyzed separately from treated participants.
Groups:
- Main Analysis Set: Participants with chronic hepatitis C (CHC) treated with pegylated interferon (peginterferon) alfa-2a monotherapy, or with peginterferon alfa-2a and ribavirin with or without other approved CHC therapy were observed. Treatments were administered according to their corresponding summary of product characteristics (SmPC).
- Elastography Analysis Set: Treated: Participants with CHC treated with peginterferon alfa-2a monotherapy, or with peginterferon alfa-2a and ribavirin with or without other approved CHC therapy were observed. The elastography analysis set includes participants, who underwent elastography and were documented in the fibroscan module. The treated set included those who were treated with hepatitis C virus (HCV) treatment as indicated.
- Elastography Analysis Set: Untreated: The untreated elastography analysis set includes those participants with CHC, who underwent elastography, were documented in the fibroscan module and were not treated with HCV treatment.
Period: Overall Study
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated | Elastography Analysis Set: Untreated
Started | 9620 | 90 | 518
Completed | 7071 | 50 | 518
Not Completed | 2549 | 40 | 0
Not completed — Patient Died | 19 | 0 | 0
Not completed — Lack of Tolerability | 305 | 3 | 0
Not completed — Lack of Virological Response | 1044 | 8 | 0
Not completed — Concomitant Disease | 74 | 2 | 0
Not completed — Lack of Compliance | 211 | 7 | 0
Not completed — Patients Request | 307 | 9 | 0
Not completed — Lost to Follow-up | 451 | 8 | 0
Not completed — Unplanned Event | 82 | 2 | 0
Not completed — Change of Laboratory Parameter | 10 | 0 | 0
Not completed — Hospitalization/Surgical Intervention | 6 | 0 | 0
Not completed — Relocation/Change of Physician | 40 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Main Analysis Set: Participants with CHC treated with peginterferon alfa-2a monotherapy, or with peginterferon alfa-2a and ribavirin with or without other approved CHC therapy were observed. Treatments were administered according to their corresponding SmPC.
- Elastography Analysis Set: Treated: Participants with CHC treated with peginterferon alfa-2a monotherapy, or with peginterferon alfa-2a and ribavirin with or without other approved CHC therapy were observed. The elastography analysis set includes participants, who underwent elastography and were documented in the fibroscan module. The treated set included those who were treated with HCV treatment as indicated.
- Total: Total of all reporting groups
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated | Elastography Analysis Set: Untreated | Total
Number analyzed (Participants) | 9620 | 90 | 518 | 10228
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.4) | 44.9 (10.5) | 51.1 (12.8) | 42.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3273 | 23 | 217 | 3513
  Male | 6347 | 67 | 301 | 6715
Number of Participants With Each Hepatitis C Viral Genotype [Number; unit: participants]
  Genotype 1 | 5699 | 51 | 377 | 6127
  Genotype 2 | 544 | 3 | 11 | 558
  Genotype 3 | 2903 | 30 | 89 | 3022
  Genotype 4 | 421 | 6 | 18 | 445
  Genotype 5 | 17 | 0 | 2 | 19
  Genotype 6 | 15 | 0 | 1 | 16
  Genotype unknown | 21 | 0 | 20 | 41
Number of Participants With Low or High Viral Load [Number; unit: participants] — Low viral load was defined as </=1,000,000 copies/milliliter (copies/ml) or </=400,000 international units/milliliter (IU/ml). High viral load was defined as >1,000,000 copies/ml or >400,000 IU/ml.
  participants
    Low viral load | 3769 | 24 | 139 | 3932
    High viral load | 5771 | 66 | 356 | 6193
    Not determined/not assessable | 80 | 0 | 23 | 103

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: RVR is defined as Hepatitis C-Virus (HCV) Polymerase Chain Reaction (PCR) assay result qualitatively negative and/or viral load ≤50 International Units/milliliter (IU/ml) at Week 4.
Time Frame: At Week 4
Population: Only treated participants were analyzed for this Outcome Measure. In each analysis set only those participants were included for whom a valid HCV PCR result was available or who discontinued from treatment before Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 6442 | 60
percentage of participants | 40.0 | 41.7

2. Primary Outcome: Percentage of Participants With Early Virologic Response (EVR)
Description: EVR is defined as HCV-PCR assay result qualitatively negative and/or decline of viral load of ≥2 log levels and/or viral load ≤50 IU/ml at Week 12.
Time Frame: At Week 12
Population: Only treated participants were analyzed for this Outcome Measure. In each analysis set only those participants were included for whom a valid HCV PCR result was available or who discontinued from treatment before Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 7383 | 54
percentage of participants | 71.2 | 77.8

3. Primary Outcome: Percentage of Participants With End of Treatment (EOT) Response
Description: EOT Response is defined as HCV-PCR assay result below limit of detection or viral load ≤50 IU/ml and/or qualitatively negative at the end of treatment.
Time Frame: Up to Week 72
Population: Only treated participants were analyzed for this Outcome Measure. All participants within each analysis set were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 9620 | 90
percentage of participants | 59.2 | 51.1

4. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR)
Description: SVR is defined as HCV-PCR assay result below limit of detection or viral load ≤50 IU/ml and/or qualitatively negative at least 12 weeks after the end of treatment at follow up. Follow-up visit occurred at 12 to 24 weeks following discontinuation of treatment.
Time Frame: Up to Week 96
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 9620 | 90
percentage of participants | 41.4 | 36.7

5. Primary Outcome: Percentage of Participants With Serious Adverse Drug Reactions (SADR)
Time Frame: Up to Week 96
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 9620 | 90
percentage of participants | 3.5 | 3.3

6. Secondary Outcome: Percentage Cumulative Dose of Peginterferon Alfa-2a Received
Description: Data for the accumulation of the cumulative dose of peginterferon alfa-2a were analyzed and reported as the percentage of the intended dose participants received. Cumulative doses were evaluated for participants for whom dosage data were documented consistently throughout the observational period. If the treatment was ongoing at the study end, the cumulative dose was aggregated for the documented observational period.
Time Frame: Up to Week 96
Population: Only treated participants were analyzed for this Outcome Measure. Only participants with evaluable data for this Outcome Measure were included in the analysis.
Measure: Median (Full Range); unit: percentage of cumulated dose
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 9005 | 90
percentage of cumulated dose | 97.9 [1.04 to 400.00] | 94.8 [4.17 to 350.00]

7. Secondary Outcome: Percentage Cumulative Dose of Ribavirin Received
Description: Data for the accumulation of the cumulative dose of ribavirin were analyzed and reported as the percentage of the intended dose participants received. Cumulative doses were evaluated for participants for whom dosage data were documented consistently throughout the observational period. If the treatment was ongoing at the study end, the cumulative dose was aggregated for the documented observational period.
Time Frame: Up to Week 96
Population: as for outcome 6
Measure: Median (Full Range); unit: percentage of cumulated dose
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 8971 | 89
percentage of cumulated dose | 100.00 [0.00 to 500.00] | 97.92 [8.33 to 480.21]

8. Secondary Outcome: Duration of Peginterferon Alfa-2a Therapy
Description: Treatment duration was evaluated for participants for whom dates of treatment start and end of therapy were documented.
Time Frame: Up to Week 72
Population: as for outcome 6
Measure: Median (Full Range); unit: weeks
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated
Number analyzed (Participants) | 8993 | 90
weeks | 27.3 [1.0 to 106.1] | 29.3 [1.1 to 84.1]

9. Secondary Outcome: Percentage of Participants With the Most Frequent Concomitant Medications
Description: Most frequent concomitant medications were defined as those, which were observed in >1 % of participants.
Time Frame: At Baseline (Day 1)
Population: Only main analysis set had evaluable data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Main Analysis Set
Number analyzed (Participants) | 9620
percentage of participants
  Anilides | 10.6
  Selective serotonin reuptake inhibitors | 9.9
  Proton pump inhibitors | 5.3
  Propionic acid derivatives | 4.7
  Propulsives | 2.3
  Other antidepressants | 2.3
  Angiotensin-converting-enzyme (ACE) inhibitors | 2.0
  Thyroid hormones | 1.8
  Corticosteroids, potent (group III) | 1.7
  Benzodiazepine related drugs | 1.5
  Pyrazolones | 1.4
  Beta blocking agents, selective | 1.3
  Non-selective monoamine reuptake inhibitors | 1.2

ADVERSE EVENTS:
Time Frame: Up to Week 96
Description: The assessment type for the Main analysis set and Elastography analysis set: treated was systematic (reported by the participants in response to questioning in the course of each study visit) whereas the assessment type for the Elastography analysis set: untreated was non-systematic (spontaneously reported by the participant).
Groups:
- Elastography Analysis Set: Treated: Participants with CHC treated with peginterferon alfa-2a monotherapy, or with peginterferon alfa-2a and ribavirin with or without other approved CHC therapy were observed. The elastography analysis set includes participants, who underwent elastography and were documented in the fibroscan module. The treated set included those, who were treated with HCV treatment as indicated.
- Elastography Analysis Set: Untreated: Participants with CHC in the untreated elastography analysis set includes those participants, who underwent elastography, were documented in the fibroscan module and were not treated with HCV treatment.
Arm/Group | Main Analysis Set | Elastography Analysis Set: Treated | Elastography Analysis Set: Untreated
Serious Adverse Events (participants affected / at risk) | 439/9620 | 4/90 | 0/518
Other Adverse Events (participants affected / at risk) | 5721/9620 | 82/90 | 0/518
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Analysis Set (N=9620) | Elastography Analysis Set: Treated (N=90) | Elastography Analysis Set: Untreated (N=518)
Anaemia (Blood and lymphatic system disorders) | 35 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Granulocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 6 | 0 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 14 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 8 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac perforation (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 3 | 0 | 0
Myocardial infarction (Cardiac disorders) | 5 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Factor VIII deficiency (Congenital, familial and genetic disorders) | 1 | 0 | 0
Intestinal atresia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 2 | 0 | 0
Ossicle disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 2 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 4 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 3 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 4 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Teeth brittle (Gastrointestinal disorders) | 1 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Asthenia (General disorders) | 3 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Death (General disorders) | 4 | 0 | 0
Disease progression (General disorders) | 1 | 0 | 0
Drug ineffective (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 0
General physical health deterioration (General disorders) | 5 | 0 | 0
Generalised oedema (General disorders) | 2 | 0 | 0
Granuloma (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0
No therapeutic response (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 8 | 0 | 0
Serositis (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 2 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 3 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0
Hepatic artery occlusion (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 3 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 5 | 0 | 0
Decreased immune responsiveness (Immune system disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 3 | 0 | 0
Abscess (Infections and infestations) | 3 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 2 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Groin abscess (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
HIV infection (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 6 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0
Nasal vestibulitis (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 27 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 6 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 5 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 2 | 0 | 0
Accident at home (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 6 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0
Biopsy liver (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 0 | 0
Blood cholinesterase decreased (Investigations) | 1 | 0 | 0
Blood count abnormal (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood glucose fluctuation (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 0
Haemoglobin decreased (Investigations) | 17 | 0 | 0
Heart rate increased (Investigations) | 1 | 0 | 0
Hepatitis C RNA increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Prothrombin time prolonged (Investigations) | 2 | 0 | 0
Renal function test abnormal (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 2 | 0 | 0
Viral load increased (Investigations) | 1 | 0 | 0
Waist circumference increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bursa disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Muscle oedema (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm malignant resectable (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 2 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 0 | 0
Hemianopia (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 4 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0
Acute psychosis (Psychiatric disorders) | 2 | 0 | 0
Aggression (Psychiatric disorders) | 2 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0
Alcohol problem (Psychiatric disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 10 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Completed suicide (Psychiatric disorders) | 3 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Dependence (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 20 | 0 | 0
Drug dependence (Psychiatric disorders) | 8 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 17 | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 0
Suicide attempt (Psychiatric disorders) | 5 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 3 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Breast induration (Reproductive system and breast disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Scrotal ulcer (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Drug abuse (Social circumstances) | 3 | 0 | 0
Drug abuser (Social circumstances) | 1 | 0 | 0
Substance use (Social circumstances) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0 | 0
Detoxification (Surgical and medical procedures) | 1 | 0 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0
Liver transplant (Surgical and medical procedures) | 0 | 1 | 0
Oophorectomy (Surgical and medical procedures) | 1 | 0 | 0
Angiodysplasia (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 0 | 0
Femoral artery embolism (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 2 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Analysis Set (N=9620) | Elastography Analysis Set: Treated (N=90) | Elastography Analysis Set: Untreated (N=518)
Anaemia (Blood and lymphatic system disorders) | 471 | 37 | 0
Leukopenia (Blood and lymphatic system disorders) | 311 | 30 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 299 | 31 | 0
Abdominal pain (Gastrointestinal disorders) | 187 | 7 | 0
Cheilitis (Gastrointestinal disorders) | 10 | 6 | 0
Gastritis (Gastrointestinal disorders) | 28 | 6 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 121 | 5 | 0
Nausea (Gastrointestinal disorders) | 820 | 16 | 0
Vomiting (Gastrointestinal disorders) | 71 | 5 | 0
Fatigue (General disorders) | 3380 | 49 | 0
Influenza like illness (General disorders) | 433 | 6 | 0
Irritability (General disorders) | 637 | 0 | 0
Pyrexia (General disorders) | 801 | 6 | 0
Oral candidiasis (Infections and infestations) | 54 | 6 | 0
Weight decreased (Investigations) | 890 | 22 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1258 | 7 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 873 | 9 | 0
Dizziness (Nervous system disorders) | 232 | 6 | 0
Headache (Nervous system disorders) | 1348 | 15 | 0
Visual field defect (Nervous system disorders) | 4 | 5 | 0
Depressed mood (Psychiatric disorders) | 865 | 16 | 0
Depression (Psychiatric disorders) | 705 | 18 | 0
Insomnia (Psychiatric disorders) | 857 | 9 | 0
Sleep disorder (Psychiatric disorders) | 234 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 247 | 12 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 555 | 6 | 0
Eczema (Skin and subcutaneous tissue disorders) | 62 | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 569 | 10 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1316 | 19 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.